CLINICAL TRIAL: NCT04829760
Title: The Effect of Psyllium and Wheat Bran on Body Weight in People With Parkinson's Disease and Constipation Symptoms
Acronym: NRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB202100363
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
Keywords: Nutrition; Dietetics; Fiber; Weight loss; Constipation; Malnutrition; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Weight Loss; Constipation; Malnutrition | interventions — Psyllium; maltodextrin

STUDY DESIGN:
Intervention Model Description: A randomized, single-blind, placebo-controlled parallel study in which participants consume 10 grams of psyllium, coarse wheat bran, or a placebo (maltodextrin) for eight weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psyllium (Experimental): 10 g per day. Participants will be instructed to divide the 10 g into 2 doses and ingest by adding the product to at least 8 ounces (240 mL) of cold water or a beverage that is typically consumed. Participants will ingest the intervention each morning and evening for eight weeks.
  Interventions: Dietary Supplement: Psyllium
- Coarse wheat bran (Experimental): 10 g per day. Participants will be instructed to divide the 10 g into 2 doses and ingest by adding the product to a food they normally eat.
  Interventions: Dietary Supplement: Coarse wheat bran
- Maltodextrin (Placebo Comparator): Volume equivalent to the psyllium. Participants will be instructed to divide the daily dose into 2 doses and ingest by adding the product to a food or to 8 ounces (240 mL) of a beverage that is typically consumed.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Psyllium — Participants will consume 10 grams of fiber from psyllium in two doses each day for 8 weeks
  Arms: Psyllium
Dietary Supplement: Coarse wheat bran — Participants will consume 10 grams of fiber from coarse wheat bran in two doses each day for 8 weeks
  Arms: Coarse wheat bran
Dietary Supplement: Maltodextrin — Participants will consume maltodextrin in a volume equivalent to the psyllium intervention (~2 tablespoons) in two doses each day for 8 weeks
  Arms: Maltodextrin

SUMMARY:
This is a 10-week randomized, controlled study to compare the safety and efficacy of two common fiber supplements, psyllium and wheat bran in terms of changes in body weight, nutrition status, and bowel function in patients with Parkinson's Disease who have constipation symptoms. After a 2-week run-in period, participants will be randomized to receive 10 grams daily of psyllium, coarse wheat bran, or maltodextrin (placebo) for 8 weeks. Nutritional and neurological evaluations will be conducted at the beginning and end of the 8-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed Parkinson's disease
* Age 40-85 years
* Drug naïve or on stable dosage of PD medications with no plans to change for the duration of the study protocol
* Hoehn & Yahr stage < 4 in the clinical "ON" state
* Using laxatives (Miralax, Dulcolax, sennosides, etc.) regularly over the past 1 months (≥ 2 days per week)
* Complete informed consent in English
* Maintain habitual diet and exercise routine throughout study period
* Consume the study intervention twice per day during the eight-week intervention period
* Complete daily and weekly questionnaires, and all dietary recalls over approximately 10 weeks
* Fast (no food or drink, except plain water, coffee, or tea) at least 12 hours before each study visit

Exclusion Criteria:

* Atypical or secondary Parkinsonism
* Underweight (BMI <18.5)
* Inability to swallow study supplement due to swallowing concerns
* Currently using a fiber supplement
* Use of another investigational product within 3 months of the screening visit
* Being treated for a physician-diagnosed GI disease or condition other than constipation, gastroparesis, gastroesophageal reflux disease, or diverticular disease

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Body weight | 8 weeks
  The difference between in mean change (final - baseline) in body weight for psyllium, wheat bran, and placebo interventions.

SECONDARY OUTCOMES:
Digestive health | Each week up to 10 weeks
  Weekly GI symptoms assessed using the Gastrointestinal Symptom Rating Scale, which is composed of 15 questions related to 5 syndromes: constipation, diarrhea, reflux, abdominal pain, and indigestion. Individual syndrome scores will be summed for a total score.
Laxative use | Each week up to 10 weeks
  Compare laxative use frequency and dosage between groups
Stool frequency | Each week up to 10 weeks
  Compare the number of stools per week between groups
Stool consistency | Each day up to 10 weeks
  Compare stool consistency, as measured by the Bristol Stool Form Scale, between groups
Body composition | 8 weeks
  Changes in muscle, fat mass, and total body water assessed by bioelectrical impedance spectroscopy.
Appetite | Each week up to 10 weeks
  Changes in appetite will be assessed weekly using the Council on Nutrition Appetite Questionnaire (CNAQ).
Nutrition risk | 8 weeks
  Changes in nutrition risk determined by the Patient Generated- Subjective Global Assessment (PG-SGA). The PG-SGA is a tool that helps clinicians determine nutrition risk by considering weight changes, changes in dietary intake, presence of nutrition impact symptoms, physical activity, comorbidities, metabolic demands, and an assessment of lean mass, fat mass, and edema.
Constipation-related Quality of Life | 8 weeks
  Changes in quality of life related to constipation assessed by the Patient Assessment of Constipation- Quality of Life questionnaire.
Non-motor symptoms | 8 weeks
  Compare non-motor symptom severity and frequency over the past 1 month will be captured by the Non-Motor Symptom Scale for Parkinson's Disease (NMSS).
Parkinson's Disease- related Quality of life | 8 weeks
  Changes in quality of life assessed by the Parkinson's disease Questionnaire 39 (PDQ-39). The PDQ-39 is a 39 questionnaire tool that assesses quality of life within the domains of activities of daily living, attention and working memory, cognition, communication, depression, functional mobility, quality of life, social relationships, and social support.
Handgrip strength | 8 weeks
  Changes in upper body strength assessed by handgrip strength via dynamometer

OTHER OUTCOMES:
Digestion-related Quality of Life | Each week up to 10 weeks
  Changes in quality of life related to digestion assessed by the Digestion-associated Quality of life Questionnaire.
Stress | Each day up to 10 weeks
  Changes in daily stress rating on a 10-point severity Likert scale.
Physical Activity | 8 weeks
  Changes in physical activity assessed by the International Physical Activity Questionnaire (IPAQ). The IPAQ assess the intensity of physical activity and sitting time to estimate total physical activity (Metabolic Equivalents-min/week).

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No